CLINICAL TRIAL: NCT05501418
Title: A Seamless Phase I/IIa Clinical Study to Evaluate the Safety and Efficacy of Allogeneic Umbilical Cord Mesenchymal Stem Cells in Patients With Severe and Critical COVID-19 Condition
Brief Title: Evaluate the Safety and Efficacy of Allogeneic Umbilical Cord Mesenchymal Stem Cells in Patients With COVID-19
Acronym: UMSC01
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ever Supreme Bio Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ES-CMSC01-C1101
Record Dates: First submitted 2022-08-10; First posted 2022-08-15 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-02

CONDITIONS: COVID-19 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- UMSC01 (Experimental): UMSC01 cells mixed with normal saline will be administered to patients after COVID-19 infection.
  Interventions: Biological: Allogeneic umbilical cord mesenchymal stem cells
- Placebo (Placebo Comparator): Normal saline will be administered to patients after COVID-19 infection.
  Interventions: Biological: Controlled normal saline

INTERVENTIONS:
Biological: Allogeneic umbilical cord mesenchymal stem cells — UMSC01 cells will be IV infusion with 12 months of follow up after treatment.
  Arms: UMSC01
Biological: Controlled normal saline — Normal saline will be IV infusion with 12 months of follow up after treatment.
  Arms: Placebo

SUMMARY:
This study is to explore the safety and efficacy of using UCMSC01 in patients with COVID-19 infection via IV stem cell administration. The novelty of the current UMSC01 treatment is the single IV infusion of UMSC01 to the worldwide emergency outbreaks of COVID-19. We hypothesize that sufficient UMSC01 retention in lung may modulate the systemic inflammatory responses.

DETAILED DESCRIPTION:
The lead Phase I safety phase will further confirm the safety profile of UMSC01 in 5 COVID-19 patients each at two dose regimens and placebo.

To start the Phase IIa study, data analysis will be performed as soon as the 21-day treatment period has been completed in the three groups. With considerations of the pandemic status and clinical practice, only one of the two active treatment groups will be selected to complete the Phase IIa study, which will recruit 60 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 20 to 80 years old.
2. Hospitalized severe and critical COVID-19 patients with laboratory confirmation by reverse-transcription polymerase chain reaction (RT-PCR) from nasopharyngeal/ oropharyngeal samples collected using standardized method.
3. Pneumonia or interstitial lung damage that is confirmed by chest radiographs or computed tomography.
4. Severe COVID-19 infection which meets any one of the following: 1) dyspnea (PR ≥ 30 times/min), 2) finger oxygen saturation ≤ 93% in the room air and resting state, 3) arterial oxygen partial pressure (PaO2)/oxygen absorption concentration (FiO2) ≤ 300 mmHg, 4) pulmonary imaging which shows that the focus progress > 50% within 24-48 hours, or
5. Critically severe COVID-19 infection which meets any of the following: 1) respiratory failure treated by mechanical ventilation, 2) shock, 3) combined with other organ failure, 4) patients expected to need ICU monitoring and treatment.
6. High sensitivity C-reactive protein (hs-CRP) serum level > 4.0 mg/dL.
7. All female patients with child-bearing potential (between puberty and 2 years after menopause) should use appropriate contraception method(s) shown below, for at least 4 weeks after UMSC01 treatment and agree to maintain such contraceptive method(s) for another 4 weeks after UMSC01 treatment.

   1. Total abstinence (when this is in line with the preferred and usual lifestyle of the subject). Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
   2. Female sterilization (bilateral oophorectomy with or without hysterectomy) or tubal ligation at least 6 weeks before taking study treatment. In case of oophorectomy alone, the reproductive status of the woman should be confirmed by the hormone level assessment.
   3. Male sterilization (at least 6 months prior to screening). For female subjects in the study, the vasectomized male partner should be the sole partner for that subject.
   4. Combination of any two of the following listed methods: (d.1 + d.2 or d.1 + d.3, or d.2 + d.3):

   d.1 Use of oral, injected, or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate < 1%), such as hormone vaginal ring or transdermal hormone contraception.

   d.2 Placement of an intrauterine device (IUD) or intrauterine system (IUS). d.3 Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository.

Exclusion Criteria:

1. Pregnancy, lactation, and those who are not pregnant but did not, or unwilling to, take effective contraceptives measures 4 weeks before and after the treatment.
2. Patients with malignant tumors or other serious systemic diseases.
3. Patients with hemoglobin < 10 g, alanine aminotransferase (ALT) ≥ 5 × ULN, aspartate aminotransferase (AST) ≥ 5 × ULN, alkaline phosphatase (ALP) ≥ 5 × ULN, total bilirubin (TBILI) ≥ 2 × ULN, serum creatinine > 2.5 mg/dl, platelet counts < 100,000/μL, WBC < 3,000 cells/μL, or neutrophil counts < 1,000/μL at screening.
4. Presence of barotrauma or hemodynamic instability defined as hypotension with diastolic blood pressure < 90 mmHg or mean arterial pressure (MAP) < 70 mmHg despite fluid expansion, and vasoactive support or pneumothorax at screening.
5. Uncontrolled hypertension with systolic blood pressure > 170 mmHg and diastolic blood pressure > 100 mmHg which, in the investigator's judgment, would not make participation appropriate.
6. Recent history of (within 2 years) ischemic heart disease or cerebrovascular attack, such as myocardial infarction, unstable angina, or stroke.
7. Recent history (within 2 years) of hypercoagulable disorder, antiphospholipid syndrome, pulmonary embolism, or deep venous thrombosis.
8. Condition other than COVID-19 that is projected to limit lifespan to ≤ 1 year.
9. History of drug or alcohol abuse within the past 24 months.
10. Unwilling to commit to follow-up visits.
11. Patients who are participating in other clinical trials with an investigational product.
12. Co-infection of HIV, tuberculosis, influenza virus, adenovirus, and other respiratory infection virus.
13. Patients with other conditions that are not suitable to participate in this clinical study as determined by the investigator.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2020-08-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Two Co-Primary Efficacy Endpoints | 21 days of the treatment period
  Proportion of patients alive with sustained improvement within the 21 days of the treatment period (Proportion Analysis), which indicates the capability of UMSC01 to save more lives
Two Co-Primary Efficacy Endpoints | 21 days of the treatment period
  Time (days) to reach sustained improvement within the 21 days of the treatment period (Time-to-Event Analysis), which indicates the capability of UMSC01 to enable patients to less suffer from the disease condition.

SECONDARY OUTCOMES:
Secondary Efficacy Endpoints | 21 days of the treatment period
  Proportion of enrolled patients alive on Day 21
Secondary Efficacy Endpoints | 21 days of the treatment period
  Proportion of enrolled patients alive and free of respiratory failure on Day 21
Secondary Efficacy Endpoints | 21 days of the treatment period
  Improvement of COVID 19 pneumonia confirmed by chest radiographs or computed tomography on Day 21 or on the day of discharge compared with baseline
Secondary Efficacy Endpoints | 21 days of the treatment period
  Improvement of clinical symptoms including duration of fever in degrees C and respiratory failure on Day 21 or on the day of discharge compared with baseline
Secondary Efficacy Endpoints | 21 days of the treatment period
  Duration of ventilator usage or oxygen therapy on Day 21 or on the day of discharge compared with baseline
Secondary Efficacy Endpoints | 21 days of the treatment period
  Levels of tumor necrosis factor-alpha (TNF-α) in pg/ml, interleukin-6 (IL-6) in pg/ml and interleukin-10 (IL-10) in pg/ml, and C-reactive protein (hsCRP) in mg/dl on Day 21 or on the day of discharge compared to baseline
Secondary Efficacy Endpoints | 21 days of the treatment period
  Troponin I level as assessed via serum blood samples on Day 21 or on the day of discharge compared with baseline
Secondary Efficacy Endpoints | 21 days of the treatment period
  ICU admission rate on Day 21 or on the day of discharge with historical data
Secondary Efficacy Endpoints | 14 days of the treatment period
  Percentage of subjects recorded in each severity rating based on Clinical classification of the COVID-19 (NCOSS scores from 1 to 8；higher scores mean a worse outcome) on Day 14 compared with historical data
Secondary Efficacy Endpoints | 21 days of the treatment period
  Percentage of subjects recorded in each severity rating based on Clinical classification of the COVID-19 (NCOSS scores from 1 to 8；higher scores mean a worse outcome) on Day 21 compared with historical data
Secondary Efficacy Endpoints | through study completion, an average of 1 year
  Average time (days) for which the patients are alive and free of respiratory failure during the treatment period
Secondary Efficacy Endpoints | 21 days of the treatment period
  Proportion of patients who need ICU care on Day 21 based on the clinical indicative of admission to ICU
Secondary Efficacy Endpoints | 21 days of the treatment period
  Proportion of patients who has been discharged form hospital on Day 21
Secondary Safety Endpoints | 21 days of the treatment period
  Number of Participants with infusion-related and allergic reactions during the treatment period
Secondary Safety Endpoints | through study completion, an average of 1 year
  Secondary infection, treatment emergent adverse event (TEAE), serious adverse event (SAE), and suspected and unexpected serious adverse reaction (SUSAR) incidences over the study period. The toxicities will be assessed by CTCAE V5.0 during the whole study period (380 days)

CONTACTS AND LOCATIONS:
Overall Officials: Woei C Shyu, Study Director — Ever Supreme Bio Technology Co., Ltd.; Long Bin Jeng, Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Non-US, Taiwan